CLINICAL TRIAL: NCT07049614
Title: Comparative Study of Postoperative Surgical Site Infections in Diabetic and Non-Diabetic Patients Undergoing General Surgical Procedures
Brief Title: Comparative Study of Postoperative Surgical Site Infections in Diabetic and Non-Diabetic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/913
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Patients
  Interventions: Diagnostic Test: Diabetic Patients
- Non-Diabetic Patients
  Interventions: Diagnostic Test: Non-Diabetic Patients

INTERVENTIONS:
Diagnostic Test: Diabetic Patients — This group consists of 66 adult diabetic patients (Type 1 or Type 2) undergoing elective general surgical procedures. These patients will be managed as per standard clinical protocols, including preoperative evaluation, glycemic control assessment (via recent HbA1c and blood glucose levels), and administration of prophylactic broad-spectrum antibiotics-typically second-generation cephalosporins and metronidazole.
  Postoperative follow-up will be conducted on Day 1, Day 7, and Day 14 to monitor for the development of surgical site infections (SSIs), which will be classified by the unit chief as superficial, deep, or organ/space infections.
  Groups: Diabetic Patients
Diagnostic Test: Non-Diabetic Patients — This group includes 66 adult non-diabetic patients undergoing elective general surgical procedures at DHQ Hospital, Dera Ismail Khan. These participants will serve as the comparison group for evaluating the incidence and characteristics of postoperative surgical site infections (SSIs). All patients will receive standard preoperative assessments and prophylactic antibiotics (second-generation cephalosporins with metronidazole) as per institutional protocols. Postoperative follow-up will be carried out on Day 1, Day 7, and Day 14, and SSIs, if any, will be classified based on CDC criteria into superficial, deep, or organ/space infections
  Groups: Non-Diabetic Patients

SUMMARY:
This prospective observational study aims to compare the incidence and characteristics of postoperative surgical site infections (SSIs) between diabetic and non-diabetic patients undergoing elective general surgical procedures.

DETAILED DESCRIPTION:
Diabetes mellitus is a well-known risk factor for delayed wound healing and postoperative complications. The study seeks to identify how diabetic status influences SSI rates, types (superficial, deep, organ/space), and associated risk factors such as glycemic control (HbA1c), duration of diabetes, and presence of comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients aged 18 to 80 years.
* Patients undergoing elective general surgical procedures.
* Patients diagnosed with diabetes mellitus (Type 1 or Type 2), whether on oral hypoglycemics or insulin, with satisfactory preoperative glycemic control.
* Patients willing to give informed consent.
* Patients available for postoperative follow-up on Day 1, 7, and 14.

Exclusion Criteria:

* Emergency surgical cases.
* Patients with gestational diabetes.
* Patients with poorly controlled diabetes preoperatively.
* Patients with severe comorbid conditions, such as ischemic heart disease, peripheral vascular disease, neuropathy, active cancer, or immunocompromised states (e.g., HIV/AIDS).
* Patients on immunosuppressive therapy.
* Patients below 18 years of age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study aims to compare the incidence and characteristics of postoperative surgical site infections (SSIs) between diabetic and non-diabetic patients undergoing elective general surgical procedures. Diabetes mellitus is a well-known risk factor for delayed wound healing and postoperative complications
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self administered questioner for data | 12 Months
  A structured questionnaire developed for this study will record demographic data (age, gender, BMI), medical history (diabetes status, duration, HbA1c levels, comorbidities), lifestyle factors (smoking status), surgical details (type of surgery, surgical approach, duration of surgery), and postoperative outcomes (SSI presence, type, day of onset, management).
  Scoring/Recording:
  Diabetes status: Diabetic / Non-Diabetic HbA1c Level: Recorded as a percentage (%) Presence of SSI: Yes / No
  Type of SSI:
  Superficial Incisional SSI. Deep Incisional SSI. Organ/Space SSI. Postoperative Complications: Sepsis, wound dehiscence, organ dysfunction (marked Yes/No).
  Hospital stay: Recorded in number of days.

CONTACTS AND LOCATIONS:
Locations (1):
- DHQ Hospital, Dera Ismāīl Khān, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No